CLINICAL TRIAL: NCT06658119
Title: Clinical Evaluation of Extended Depth-of-focus Intraocular Lens in Refractive Cataract Surgery
Brief Title: Clinical Evaluation of Extended Depth-of-focus Intraocular Lens in Refractive Cataract Surgery: a Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20241068
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-10

CONDITIONS: Cataract
Keywords: cataract surgery; intraocular lens; extended depth-of-focus
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction; Lens Implantation, Intraocular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tecnis Synergy ZFR00 IOL (Experimental): Tecnis Synergy ZFR00 IOL will be implanted in the patient's eye during cataract surgery.
  Interventions: Procedure: cataract surgery
- Tecnis Symfony ZXR00 IOL (Placebo Comparator): Tecnis Symfony ZXR00 IOL will be implanted in the patient's eye during cataract surgery.
  Interventions: Procedure: cataract surgery

INTERVENTIONS:
Procedure: cataract surgery — The participants will receive femtosecond laser-assisted cataract surgery and implant an extended depth-of-focus intraocular lens (Tecnis Synergy ZFR00).
  Other Names: intraocular lens implantation
  Arms: Tecnis Synergy ZFR00 IOL
Procedure: cataract surgery — The participants will receive femtosecond laser-assisted cataract surgery and implant an extended depth-of-focus intraocular lens (Tecnis Symfony ZXR00).
  Other Names: intraocular lens implantation
  Arms: Tecnis Symfony ZXR00 IOL

SUMMARY:
The goal of this clinical trial is to compare the clinical outcomes of two extended depth-of-focus intraocular lens after cataract surgery. The randomized controlled trail will enroll 90 participants. The participants will be randomly assigned to implant Tecnis Synergy ZFR00 or Tecnis Symfony ZXR00 intraocular lens. Follow-up visit will be performed till 3 months postoperatively to compare the visual acuity, subjective manifest refraction, and visual quality between groups.

ELIGIBILITY:
Inclusion Criteria:

* age-related cataract patients aged between 40 to 80
* patients with preoperative astigmatism less than 0.75 D, and kappa value less than 0.7 mm
* patients who plan to receive femtosecond laser-assisted cataract surgery

Exclusion Criteria:

* patients with ocular surface abnormalities such as irregular corneal astigmatism, corneal scarring, keratoconus, and pterygium)
* patients with history of ocular trauma or surgery
* patients with coexisting ocular disorders such as glaucoma, retinal vascular occlusive disease, retinal detachment, diabetic retinopathy, and any optic nerve-related pathologies
* patients with concurrent severe systemic diseases
* patients who lack of cooperation

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | 1 day, 1 week, 1 month, 3 months postoperatively
  Visual acuity will be assessed using the Standard Logarithmic Visual Acuity Chart. The results will be recorded in decimal and converted to logMAR and Snellen equivalent.

SECONDARY OUTCOMES:
Visual quality | 3 months postoperatively
  OPD-scan measurement. Higher-order aberration, tilt and decentration will be recorded.
defocus curve | 3 months postoperatively
  Best distance visual acuity varied from - 5.00 to + 2.00 D in steps of 0.50 D under photopic conditions was recorded.
contrast sensitivity | 3 months postoperatively
  Contrast sensitivity will be converted to logarithmic scale before analysis and referred to as log-contrast sensitivity.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Center of the Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.